CLINICAL TRIAL: NCT05983536
Title: The Evaluation of Anti-interference Ability and Clinical Specificity of HIV Ag +Ab Assay Kit (Sysmex)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 89269678
Record Dates: First submitted 2023-07-18; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: HIV Seropositivity; Cancer; Blood Disease
MeSH Terms: conditions — HIV Seropositivity; Neoplasms; Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer patients: Cancer patints that confirmed by pathological examination
  Interventions: Diagnostic Test: HIV Ag +Ab Assay Kit (Sysmex)
- Patients with blood diseases: Bone marrow aspiration and biopsy confirmed the blood disease
  Interventions: Diagnostic Test: HIV Ag +Ab Assay Kit (Sysmex)

INTERVENTIONS:
Diagnostic Test: HIV Ag +Ab Assay Kit (Sysmex) — Using the HIV Ag +Ab Assay Kit (Sysmex) to detect the HIV antigen and antibody in serum, then verified by Human Immunodeficiency Virus (HIV 1+2) Antibody Test Kit (Immunoimprinting). The specificity of the HIV Ag +Ab Assay Kit (Sysmex) is calculated according to the specificity calculation formula.

SUMMARY:
To evaluate the anti-interference and specificity of HIV Ag +Ab Assay Kit (Sysmex) for the detection of HIV antigens and antibodies.

DETAILED DESCRIPTION:
First,HIV Ag +Ab Assay Kit (Sysmex)Assay Kit (Sysmex) was used to detect HIV antigens and antibodies in the serum of patients with tumor and blood diseases, and then confirmed by using the gold standard for HIV diagnosis,human immunodeficiency virus (HIV type 1+2) antibody assay kit (immunoimprinting). The specificity of HIV Ag +Ab Assay Kit (Sysmex) for HIV assay in patients with tumor and hematological diseases was calculated.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of tumor Disease or blood disease
* Blood samples must meet the test requirements

Exclusion Criteria:

* N/A

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients and blood disease patients with age over 18 and have an HIV test in that very day.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-09-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
The HIV Ab/Ag results | through study completion, an average of 1.5 year
  The HIV Ab/Ag results generated using HIV Ag +Ab Assay Kit (Sysmex) and the gold standard method for HIV test. The results will be recoreded seperately.

CONTACTS AND LOCATIONS:
Overall Officials: Xia Zhao, Master, Principal Investigator — Qianfoshan Hospital

IPD SHARING:
Plan to Share IPD: Undecided
The planed will be shared after the clinical trial is completed and the patent protection is obtained

REFERENCES:
- [Background] Alali M, Carlucci JG, Christenson J, Prather C, Skiles J. Case Series of False-Positive HIV Test Results in Pediatric Acute Lymphoblastic Leukemia Patients Following Chimeric Antigen Receptor T-Cell Therapy: Guidance on How to Avoid and Resolve Diagnostic Dilemmas. J Pediatric Infect Dis Soc. 2022 Aug 30;11(8):383-385. doi: 10.1093/jpids/piac028. PMID 35512447
- [Background] Lu X, Zhang M, Liu W, Sheng N, Du Q, Zhang M, Guo X, Wang G, Wang Q. A method to alleviate false-positive results of the Elecsys HIV combi PT assay. Sci Rep. 2021 Jan 13;11(1):1033. doi: 10.1038/s41598-020-80047-0. PMID 33441741